CLINICAL TRIAL: NCT02620865
Title: Phase Ib/II Treatment of Advanced Pancreatic Cancer With Anti-CD3 x Anti-EGFR-Bispecific Antibody Armed Activated T-Cells (BATs) in Combination With Low Dose IL-2 and GM-CSF
Brief Title: BATS With in Combination With Low Dose IL-1 and GM-CSF for Advanced Pancreatic Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Barbara Ann Karmanos Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Anthony F. Shields, MD PhD, Principal Investigator, Barbara Ann Karmanos Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015-100; NCI-2015-01942 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2015-100 (Other: Wayne State University/Karmanos Cancer Institute); P30CA022453 (NIH)
Record Dates: First submitted 2015-12-01; First posted 2015-12-03 (Estimated); Results first posted 2023-05-15 (Actual); Last update posted 2023-05-15 (Actual); Status verified 2023-04

CONDITIONS: Metastatic Pancreatic Adenocarcinoma; Recurrent Pancreatic Carcinoma; Stage III Pancreatic Cancer; Stage IV Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — aldesleukin; Immunization, Passive; Fluorouracil; dehydroftorafur; Gemcitabine; Irinotecan; Leucovorin; Oxaliplatin; Taxes; Albumin-Bound Paclitaxel; 130-nm albumin-bound paclitaxel; sargramostim; Colony-Stimulating Factors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (anti-CD3 x anti-EGFR BATs) (Experimental): Patients receive one of the following standard chemotherapy regimens at the discretion of the treating physician: gemcitabine hydrochloride IV over 30 minutes; gemcitabine hydrochloride IV over 30 minutes and paclitaxel albumin-stabilized nanoparticle formulation IV over 30-40 minutes; oxaliplatin IV over 2 hours, fluorouracil IV over 46 hours and leucovorin calcium IV over 2 hours; or fluorouracil IV over 46 hours, leucovorin calcium IV over 2 hours, irinotecan hydrochloride IV, and oxaliplatin IV over 2 hours. Approximately 2 weeks after standard chemotherapy completion, patients receive anti-CD3 x anti-EGFR-bispecific antibody armed activated T-cells IV over 5-30 minutes twice weekly for 4 weeks. Patients also receive aldesleukin SC and sargramostim SC on day -3 before the first anti-CD3 x anti-EGFR-bispecific antibody armed activated T-cells infusion and continuing twice weekly until the final infusion.
  Interventions: Biological: Aldesleukin; Biological: Antibody Therapy; Drug: Fluorouracil; Drug: Gemcitabine Hydrochloride; Drug: Irinotecan Hydrochloride; Other: Laboratory Biomarker Analysis; Drug: Leucovorin Calcium; Drug: Oxaliplatin; Drug: Paclitaxel Albumin-Stabilized Nanoparticle Formulation; Biological: Sargramostim

INTERVENTIONS:
Biological: Aldesleukin — Given SC
  Other Names: 125-L-Serine-2-133-interleukin 2; Proleukin; r-serHuIL-2; Recombinant Human IL-2; Recombinant Human Interleukin-2
Biological: Antibody Therapy — Given anti-CD3 x anti-EGFR-bispecific antibody armed activated T-cells IV
  Other Names: passive antibody therapy
Drug: Fluorouracil — Given IV
  Other Names: 5-Fluoro-2,4(1H, 3H)-pyrimidinedione; 5-Fluorouracil; 5-Fluracil; 5-FU; AccuSite; Actino-Hermal; Adrucil; Arumel; Cytosafe; Efudex; Efurix; Fiverocil; Fluoro Uracil; Fluoroplex; Fluouracil; Flurablastin; Fluracedyl; Fluracil; Fluril; Fluroblastin; Flurox; Ribofluor; Ro 2-9757; Ro-2-9757; Timazin
Drug: Gemcitabine Hydrochloride — Given IV
  Other Names: dFdCyd; Difluorodeoxycytidine Hydrochloride; Gemzar; LY-188011
Drug: Irinotecan Hydrochloride — Given IV
  Other Names: Campto; Camptosar; Camptothecin 11; Camptothecin-11; CPT 11; CPT-11; U-101440E
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Leucovorin Calcium — Given IV
  Other Names: Adinepar; Calcifolin; Calcium (6S)-Folinate; Calcium Folinate; Calcium Leucovorin; Calfolex; Calinat; Cehafolin; Citofolin; Citrec; Citrovorum Factor; Cromatonbic Folinico; Dalisol; Disintox; Divical; Ecofol; Emovis; Factor, Citrovorum; Flynoken A; Folaren; Folaxin; FOLI-cell; Foliben; Folidan; Folidar; Folinac; Folinate Calcium; folinic acid; Folinic Acid Calcium Salt Pentahydrate; Folinoral; Folinvit; Foliplus; Folix; Imo; Lederfolat; Lederfolin; Leucosar; leucovorin; Rescufolin; Rescuvolin; Tonofolin; Wellcovorin
Drug: Oxaliplatin — Given IV
  Other Names: 1-OHP; Dacotin; Dacplat; Diaminocyclohexane Oxalatoplatinum; Eloxatin; Eloxatine; JM-83; Oxalatoplatin; Oxalatoplatinum; RP 54780; RP-54780; SR-96669
Drug: Paclitaxel Albumin-Stabilized Nanoparticle Formulation — Given IV
  Other Names: ABI 007; ABI-007; Abraxane; Albumin-bound Paclitaxel; Albumin-Stabilized Nanoparticle Paclitaxel; nab-paclitaxel; Nanoparticle Albumin-bound Paclitaxel; Nanoparticle Paclitaxel; protein-bound paclitaxel
Biological: Sargramostim — Given SC
  Other Names: 23-L-Leucinecolony-Stimulating Factor 2; DRG-0012; Leukine; Prokine; rhu GM-CFS; Sagramostim; Sargramostatin

SUMMARY:
This phase Ib/II trial studies the side effects and best dose of bispecific antibody armed activated T-cells when given together with aldesleukin and sargramostim and to see how well they work in treating patients with pancreatic cancer that has spread from where it started to nearby tissue or lymph nodes (locally advanced) or other places in the body (metastatic). Bispecific antibody armed activated T-cells are the patient's own T cells that are coated with a bispecific antibody comprising 2 antibodies chemically joined together. These antibodies have specific targets and binding properties that may give the T cells a greater ability to seek out, attach to, and kill more cancer cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Confirm in a single dose phase I (3 to 6 patients [pts]) that 8 infusions of 10^10 epidermal growth factor receptor (EGFR) bispecific antibody armed activated T cells (BATs) given twice per week in combination with interleukin (IL)-2 (aldesleukin) (300,000 IU/m^2/day) and granulocyte-macrophage colony stimulating factor (GM-CSF) (sargramostim) (250 ug/m^2/twice weekly) beginning 3 days before the 1st infusion and ending on the day of the last infusion is safe.

II. Perform a phase II clinical trial to estimate the clinical efficacy of 8 infusions of 10^10 EGFR BATs in combination with IL-2 and GM-CSF in 39 evaluable pts (including the 3-6 pts in the single dose phase I).

SECONDARY OBJECTIVES:

I. Determine if infusions of EGFR BATs significantly increase cellular or humoral anti-pancreatic cancer (PC) responses by peripheral blood mononuclear cells (PBMC) at different time points after last EGFR BATs infusion and if those responses persist beyond 2 months (mos).

II. Obtain original tumor paraffin blocks prior to treatment and evaluate blocks for cluster of differentiation (CD)3, CD4, CD8, programmed cell death (PD)1/programmed cell death ligand (PDL)1, monocytes subpopulations, myeloid-derived suppressor cells (MDSC), and cytoplasmic interferon (IFN)-gamma and IL-10 by immunohistochemical staining to quantitate type and number of tumor infiltrating lymphocytes (TILs) in the tumor microenvironment to estimate whether the type and number correlate with clinical responses.

III. To determine the time to progression (TTP).

OUTLINE: This is a phase Ib, dose-escalation study of anti-CD3 x anti-EGFR-bispecific antibody armed activated T-cells followed by a phase II study.

Patients receive one of the following standard chemotherapy regimens at the discretion of the treating physician: gemcitabine hydrochloride intravenously (IV) over 30 minutes; gemcitabine hydrochloride IV over 30 minutes and paclitaxel albumin-stabilized nanoparticle formulation IV over 30-40 minutes; oxaliplatin IV over 2 hours, fluorouracil IV over 46 hours and leucovorin calcium IV over 2 hours; or fluorouracil IV over 46 hours, leucovorin calcium IV over 2 hours, irinotecan hydrochloride IV, and oxaliplatin IV over 2 hours. Approximately 2 weeks after standard chemotherapy completion, patients receive anti-CD3 x anti-EGFR-bispecific antibody armed activated T-cells IV over 5-30 minutes twice weekly for 4 weeks. Patients also receive aldesleukin subcutaneously (SC) and sargramostim SC on day -3 before the first anti-CD3 x anti-EGFR-bispecific antibody armed activated T-cells infusion and continuing twice weekly until the final infusion.

After completion of study treatment, patients are followed up for 18 months.

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological proof of pancreatic adenocarcinoma; must have locally advanced or metastatic pancreatic cancer who have received at least first line chemotherapy and may have responding, stable or progressive disease
* Expected survival >= 3 months
* Karnofsky performance scale (KPS) >= 70% or Southwestern Oncology Group (SWOG) performance status 0 or 1
* Absolute neutrophil count (ANC) >= 1,000/mm^3
* Lymphocyte count >= 400/mm^3
* Platelet count >= 75,000/mm^3
* Hemoglobin >= 8 g/dL
* Serum creatinine < 2.0 mg/dl, creatinine clearance >= 50 ml/mm (can be calculated or measured)
* Total bilirubin =< 2 mg/dl (biliary stent is allowed)
* Serum glutamate pyruvate transaminase (SGPT) and serum glutamic oxaloacetic transaminase (SGOT) < 5.0 times normal
* Left ventricular ejection fraction (LVEF) >= 45% at rest (multigated acquisition scan [MUGA] or echocardiogram [Echo])
* Females of childbearing potential, and males, must be willing to use an effective method of contraception
* Females of childbearing potential must have a negative pregnancy test within 7 days of being registered for protocol therapy

Exclusion Criteria:

* Any chemotherapy related toxicities from prior treatment (> grade 2 per Common Terminology Criteria for Adverse Events [CTCAE] version [v]4.0)
* Known hypersensitivity to cetuximab or other EGFR antibody
* Treatment with any investigational agent within 14 days prior to being registered for protocol therapy
* Symptomatic brain metastasis
* Chronic treatment with systemic steroids or another immuno-suppressive agent
* Serious non-healing wound, ulcer, bone fracture, major surgical procedure, open biopsy or significant traumatic injury within 28 days prior to being registered for protocol therapy
* Active liver disease such as cirrhosis, chronic active hepatitis or chronic persistent hepatitis
* Known human immunodeficiency virus (HIV) infection
* Active bleeding or a pathological condition that is associated with a high risk of bleeding (therapeutic anticoagulation is allowed)
* Has an active infection requiring systemic therapy
* A serious uncontrolled medical disorder that in the opinion of the investigator may be jeopardized by the treatment with protocol therapy
* Females must not be breastfeeding
* Patient (Pt) may be excluded if, in the opinion of the principal investigator (PI) and investigator team, the pt is not capable of being compliant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2015-12; Primary Completion 2021-06-21 (Actual); Study Completion 2021-06-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Shields, Principal Investigator — Barbara Ann Karmanos Cancer Institute
Locations (1):
- Wayne State University/Karmanos Cancer Institute, Detroit, Michigan, United States

REFERENCES:
- [Derived] Lum LG, Thakur A, Choi M, Deol A, Kondadasula V, Schalk D, Fields K, Dufrense M, Philip P, Dyson G, Aon HD, Shields AF. Clinical and immune responses to anti-CD3 x anti-EGFR bispecific antibody armed activated T cells (EGFR BATs) in pancreatic cancer patients. Oncoimmunology. 2020 Jun 10;9(1):1773201. doi: 10.1080/2162402X.2020.1773201. PMID 32939319

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Anti-CD3 x Anti-EGFR BATs)
Started | 2
Completed | 2
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Anti-CD3 x Anti-EGFR BATs)
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 1
Age, Continuous [Mean (Full Range); unit: years] | 63 [54 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: Median Overall Survival (OS)
Description: Descriptive statistics (point and exact 90% confidence interval estimates from the resultant Kaplan-Meier curve) will be generated for OS. The median OS will be estimated on an intention-to-treat basis (using all registered patients), and on a response-evaluable basis (using all patients who completed all BAT infusions) using the Kaplan-Meier method.
Time Frame: Up to 18 months
Measure: Median (90% Confidence Interval); unit: years
Arm/Group | Treatment (Anti-CD3 x Anti-EGFR BATs)
Number analyzed (Participants) | 2
years | 0.934 [0.934 to NA] — Median survival (MS) is calculated by using the Kaplan-Meier (KM) curve. The MS is found by seeing where the estimated KM curve intersects with the horizontal line indicating 50% survival (HL-50). The upper 90% confidence value for the MS is found by seeing where the upper confidence band (CB) for the KM estimate intersects with HL-50. For this analysis, the upper CB is 1 for the whole time period under study; which means that it never intersects with HL-50; and thus is not available to report

2. Secondary Outcome: Biomarker Analysis (Including CD3, CD4, CD8, PD1, PDL1, Monocytes, MDSC, IFN-gamma, IL-10, and TILs) Assessed Using Immunohistochemistry
Description: Each biomarker and computed biomarker will be evaluated for normality and transformed (including non-parametric) if necessary to achieve normality. Summary statistics (including means, medians, and standard deviations) will be produced for each variable and subsequently associate each variable with OS using Cox regression. In addition, a threshold for each variable associating with OS will be defined using classification and regression trees.
  The tumor will be stained for inflammatory biomarkers. Specifically, T cells with undergo cytoplasmic staining for IFN and IL-10 and the level and ratio of these markers will be evaluated.
Time Frame: Up to 18 months
Population: Analysis cannot be performed since data were not collected
Arm/Group | Treatment (Anti-CD3 x Anti-EGFR BATs)
Number analyzed (Participants) | 0

3. Secondary Outcome: Incidence of Toxicity (CTCAE Version 4.0)
Description: Toxicity rates will be estimated using all treated patients.
Time Frame: Up to 18 months
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Anti-CD3 x Anti-EGFR BATs)
Number analyzed (Participants) | 2
Participants
  Anorexia | 1
  Anxiety | 1
  Chills | 2
  Depression | 1
  Diarrhea | 2
  Dizziness | 1
  Dry Mouth | 1
  Fatigue | 2
  Fever | 2
  Gastroesophageal reflux disease | 1
  Headache | 2
  Myalgia | 1
  Nausea | 2
  Rash maculo-papular | 2
  Vomiting | 1

4. Secondary Outcome: Progression Free Survival (PFS)
Description: Descriptive statistics (point and exact 90% confidence interval estimates from the resultant Kaplan-Meier curve) will be generated for PFS. The median PFS will be estimated on an intention-to-treat basis (using all registered patients), and on a response-evaluable basis (using all patients who completed all BAT infusions) using the Kaplan-Meier method.
Time Frame: Up to 18 months
Measure: Median (90% Confidence Interval); unit: Years
Arm/Group | Treatment (Anti-CD3 x Anti-EGFR BATs)
Number analyzed (Participants) | 2
Years | 0.934 [0.934 to NA] — Median survival (MS) is calculated by using the Kaplan-Meier (KM) curve. The MS is found by seeing where the estimated KM curve intersects with the horizontal line indicating 50% survival (HL-50). The upper 90% confidence value for the MS is found by seeing where the upper confidence band (CB) for the KM estimate intersects with HL-50. For this analysis, the upper CB is 1 for the whole time period under study; which means that it never intersects with HL-50; and thus is not available to report

5. Secondary Outcome: Quantitative Immune Response
Description: For the quantitative immune response variables, summary statistics (including means, medians, and standard deviations) will be produced pre- and post-BATs treatment. Subsequent analyses will compare the immune response variables (after a suitable transformation, if necessary) pre- and post-treatment using a paired t-test (or Wilcoxon sign ranked test if the data are not approximately normally distributed). To explore whether immune responses associate with clinical responses, the association between the baseline of each biomarker and clinical endpoints (such as response, or OS) will be analyze
Time Frame: Up to 18 months
Population: Analysis cannot be performed since data were not collected
Arm/Group | Treatment (Anti-CD3 x Anti-EGFR BATs)
Number analyzed (Participants) | 0

6. Secondary Outcome: TTP
Description: To explore whether immune responses associate with clinical responses, the association between the baseline of each biomarker and clinical endpoints (such as response, or OS) will be analyzed using logistic regression for binary endpoints and Cox regression for time to event endpoints.
Time Frame: Up to 18 months
Population: Analysis cannot be performed since data were not collected
Arm/Group | Treatment (Anti-CD3 x Anti-EGFR BATs)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse event data was collected up to 3 months after off-treatment date, up to 18 months.
Description: The definitions do not differ.
Arm/Group | Treatment (Anti-CD3 x Anti-EGFR BATs)
All-Cause Mortality (participants affected / at risk) | 1/2
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 2/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Anti-CD3 x Anti-EGFR BATs) (N=2)
Anorexia (Gastrointestinal disorders) | 1
Anxiety (General disorders) | 1
Chills (General disorders) | 2
Depression (Psychiatric disorders) | 1
Diarrhea (Gastrointestinal disorders) | 2
Dizziness (Nervous system disorders) | 1
Dry Mouth (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 2
Fever (General disorders) | 2
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1
Headache (Nervous system disorders) | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Nausea (Gastrointestinal disorders) | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1
Vomiting (Gastrointestinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-05-27): https://cdn.clinicaltrials.gov/large-docs/65/NCT02620865/Prot_SAP_000.pdf